CLINICAL TRIAL: NCT01977157
Title: Alcohol Detection Via Bioimpedance Mesurements
Acronym: AlkBIS
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 11-189
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Impedance cardiography; bioimpedance; spectroscopy; extracellular resistance; body composition; hemodynamics; alcohol

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bioimpedance measurements while trinking alcohol: Bioimpedance spectroscopy (BIS) measurements on 12 healthy subjects were performed while they were drinking alkohol until reaching a BAC of 0.8 ‰.
  Interventions: Device: bioimpedance mesurements

INTERVENTIONS:
Device: bioimpedance mesurements — Bioimpedance measurements were conducted with a BIS device (SFB7, ImpediMed, Pinkeba, Australia) covering a frequency range between 5 kHz and 1 MHz and an ICG device (Niccomo, medis, Ilmenau, Germany)

SUMMARY:
Examination if the bioimpendanz measurement can be used for the determination of the alcohol content in human blood.

Furthermore the blood alcohol content (BAC) will be estimated by an official breathalyzer and one blood test.

DETAILED DESCRIPTION:
In this clinical trail it will be analyzed, if it is possible to assess the blood alcohol content (BAC) with the bioimpedance devices (SFB7, ImpediMed; Nicomo).

This technology is non-invasive an can be measured by using conductive electrodes, capacitive electrodes or inductive measurement systems.

The BIS-values will be compared with an official breathanalyzer (Alcotest 7110 Evidential MK III, Dräger, Lübeck, Germany).

Furthermore one blood sample will be taken and analyzed with the ADH method as the current gold standard at the end of the trail.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* able to give informed consent
* Inconspicuous laboratory and drug screening

Exclusion Criteria:

* electrophobica
* alcoholphobica, -allergy
* metallic ans / or electric implants
* underage persons
* interactively medication

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male subjects
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Bioimpedance measurements | 4 hours
  Evaluation if the bioimpedance measurements can be used to verify and quantify the alcohol content in human blood. Bioimpedance measurements will be conducted with the BIS device (SFB7, ImpediMed) covering a frequency range between 5 kHz and 1 MHz and an ICG device (Niccomo,medis) operating at. The whole-body and hand-to-hand bioimpedance will be analyzed. Extracellular resistance (Re), intracellular resistance (Ri) and capacitive effects (Cm) are calculated by using the Cole model Grimnes (2000).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Czaplik, Dr. med., Principal Investigator — Department of Anaesthesiology ,Chair for Medical Information Technology Helmholtz Institute for Biomedical Engineering RWTH Aachen University
Locations (1):
- Department of Anaesthesiology, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany